CLINICAL TRIAL: NCT03858777
Title: Cardiomyocyte Specific Cell Free DNA as a Marker of Cardiac Sarcoidosis
Brief Title: Cell Free DNA in Cardiac Sarcoidosis
Acronym: cfDNA in CS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nabeel Hamzeh (Other)
Responsible Party: Sponsor-Investigator, Nabeel Hamzeh, Associate Professor of Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201812737
Record Dates: First submitted 2019-02-25; First posted 2019-03-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Sarcoidosis With Myocarditis; Sarcoidosis; Healthy; ST Elevation Myocardial Infarction
Keywords: sarcoidosis
MeSH Terms: conditions — Sarcoidosis; ST Elevation Myocardial Infarction | interventions — Noninvasive Prenatal Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Sarcoidosis patients without evidence of active myocarditis (Active Comparator): A single blood draw.
  Interventions: Diagnostic Test: cell free DNA
- Sarcoidosis patients with evidence of active myocarditis (Experimental): Two blood draws 2 months apart.
  Interventions: Diagnostic Test: cell free DNA
- Acute ST elevation myocardial infarction (STEMI) (Active Comparator): Three blood draws, baseline, 6 hours and 24 hours.
  Interventions: Diagnostic Test: cell free DNA
- Healthy controls (Placebo Comparator): A single blood draw
  Interventions: Diagnostic Test: cell free DNA

INTERVENTIONS:
Diagnostic Test: cell free DNA — All groups will have blood draws and cfDNA measured

SUMMARY:
Sarcoidosis is a multisystem granulomatous disease of unknown cause that can affect any organ in the body, including the heart. Granulomatous myocarditis can lead to ventricular dysfunction and ventricular arrhythmias causing significant morbidity and mortality. Immunosuppressive therapy (IST) has been shown to reverse active myocarditis and preserve left ventricular (LV) function and in some cases improve LV function. In addition, IST can suppress arrhythmias that develop due to active myocarditis and prevent the formation of scar.

The potential role of cardiac biomarkers, including brain natriuretic peptide (BNP), atrial natriuretic peptide (ANP), and cardiac troponins, in detecting active myocarditis is limited and studies have been disappointing. At present, there are no biomarkers to detect active myocarditis and the use of advanced imaging modalities (FDG-PET) for assessing and monitoring active myocarditis is not feasible or practical and is associate with high radiation exposure. As such, a biomarker that is reflective of active myocarditis and that is cardiac specific will assist physicians in assessing the presence of active myocarditis to guide therapeutic decisions and to assess response to therapy which can limit further cardiac damage.

Cell free DNA (cfDNA) are fragments of genomic DNA that are released into the circulation from dying or damaged cells. It is a powerful diagnostic tool in cancer, transplant rejection and fetal medicine especially when the genomic source differs from the host. A novel technique that relies on tissue unique CpG methylation patterns can identify the tissue source of cell free DNA in an individual reflecting potential tissue injury. We will be conducting a pilot study to explore the utility of this diagnostic tool to identify granulomatous myocarditis in patients with sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystem granulomatous disease of unknown cause that can affect any organ in the body, including the heart. Sarcoidosis results from an immune reaction to an environmental exposure to yet unknown antigen(s) in a genetically predisposed individual. Autopsy studies have suggested that cardiac involvement with sarcoidosis occurs in up to 25% of cases, although more than half of these cases are sub-clinical. Cardiac sarcoidosis (CS) CS can lead to life-threatening heart failure, heart block, or rhythm disturbance and accounts for 13-25% of all sarcoidosis deaths in the USA. Therefore, although respiratory failure from lung sarcoidosis is the most common cause of sarcoidosis-related death in the USA, sudden death from cardiac sarcoidosis is a major concern owing to its acute nature. CS can present in a multitude of ways. It can be the initial manifestation of sarcoidosis in an individual not known to have sarcoidosis (a cohort beyond the aims of this proposal), patients can present with cardiac symptoms which can include palpitations, near-syncope or syncopal episodes which require a complete workup for potential CS and patients can be asymptomatic which is a sizable cohort considering the discrepancy between the expected prevalence of CS (25-40%) and CS that is detected clinically (5%).

Granulomatous myocarditis can lead to ventricular dysfunction and ventricular arrhythmias causing significant morbidity and mortality. Immunosuppressive therapy (IST) has been shown to reverse active myocarditis and preserve left ventricular (LV) function and in some cases improve LV function. In addition, IST can suppress arrhythmias that develop due to active myocarditis and prevent the formation of scar. Cardiac MRI (cMRI) and cardiac PET scans are currently used as complementary diagnostic tests for cardiac sarcoidosis, although with some limitations. Cardiac MRI with gadolinium has a sensitivity of 76-100% and specificity of 78-92% for the diagnosis of cardiac sarcoidosis, but its use is limited in patients with implantable cardiac devices. The presence of delayed enhancement on gadolinium-enhanced MRI is suggestive of scar tissue formation. 18FDG PET uses radioactive glucose to detect areas of active inflammation. The use of 18FDG PET as a marker of active granulomatous myocarditis should be interpreted carefully as several studies have shown the limitations of such protocols that force the myocardium to generate energy using free fatty acid metabolism exclusively. In addition, studies have also shown that the presumed pathological patterns, focal and focal on diffuse uptake, are also seen in healthy controls and patients with ischemic congestive heart failure who have undergone 18-FDG-PET12 and that a blood glucose level of >7.5mmol/L (>137mg/dl) at the time of the study results in absent or minimal myocardial FDG activity.

The potential role of cardiac biomarkers, including brain natriuretic peptide (BNP), atrial natriuretic peptide (ANP), and cardiac troponins, in detecting active myocarditis is limited and studies have been disappointing. At present, there are no biomarkers to detect active myocarditis and the use of advanced imaging modalities (FDG-PET) for assessing and monitoring active myocarditis is not feasible or practical and is associate with high radiation exposure. As such, a biomarker that is reflective of active myocarditis and that is cardiac specific will assist physicians in assessing the presence of active myocarditis to guide therapeutic decisions and to assess response to therapy which can limit further cardiac damage.

Cell free DNA (cfDNA) are fragments of genomic DNA that are released into the circulation from dying or damaged cells. It is a powerful diagnostic tool in cancer, transplant rejection and fetal medicine especially when the genomic source differs from the host. A novel technique that relies on tissue unique CpG methylation patterns can identify the tissue source of cell free DNA in an individual reflecting potential tissue injury. A recent paper utilized this technique to identify cardiac specific cfDNA in the bloodstream of patients with acute myocardial injury and sepsis reflecting cardiomyocyte injury/death. We will be conducting a pilot study to explore the utility of this diagnostic tool to identify granulomatous myocarditis in patients with sarcoidosis.

ELIGIBILITY:
1. Sarcoidosis patients without evidence of active myocarditis:

   * Inclusion:

     * Diagnosis of sarcoidosis based on the ATS/ERS criteria.
     * Normal 12 lead ECG within the past one year.
     * Non-smoker.
     * No immunosuppressive therapy for at least one year.
   * Exclusion:

     * Known cardiac disease.
     * Active smoker.
     * On immunosuppressive therapy.
2. Sarcoidosis patients with evidence of active myocarditis:

   * Inclusion:

     * Diagnosis of sarcoidosis based on the ATS/ERS criteria.
     * Evidence of active myocarditis based on recent cMRI or cFDG-PET.
     * Non-smoker.
   * Exclusion:

     * Known cardiac disease other than sarcoidosis.
     * Active smoker.
     * On immunosuppressive therapy.
3. Acute ST elevation myocardial infarction (STEMI):

   * Inclusion:

     * Diagnosis STEMI based on 1mm ST elevation in 2 or more contiguous leads.
     * Symptom onset within 12 hours.
     * Undergoing cardiac intervention for acute coronary syndrome.
     * Able to consent for blood draw.
   * Exclusion:

     * Active smoker.
     * Hemodynamically unstable.
4. Healthy controls:

   * Inclusion:

     * No known cardiac disease.
     * No known cardiovascular risk factors: hypertension, diabetes.
     * Non-smoker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
cfDNA level | cfDNA level at baseline and 2 months for sarcoidosis with heart disease compared to cfDNA levels at baseline for healthy controls and sarcoidosis without cardiac disease and cfDNA levels at baseline, 6 and 24 hours for STEMI patients.
  cfDNA level

CONTACTS AND LOCATIONS:
Overall Officials: Nabeel Hamzeh, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No